CLINICAL TRIAL: NCT03959410
Title: Impact of HPV on a Cohort of Southern Italian Women: a Prospective Observational Study About Epidemiological, Clinical, Morphological and Microbiological Features of HPV Infection
Brief Title: Impact of HPV on a Cohort of Southern Italian Women: Epidemiological, Clinical, Morphological and Microbiological Features
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Pasquale De Franciscis, Associate Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N.594
Record Dates: First submitted 2019-05-21; First posted 2019-05-22 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Cervix Cancer
Keywords: hpv; cervical cancer; microbiome
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HPV-positive patients (Active Comparator): Patients who are positive for HPV DNA test
  Interventions: Diagnostic Test: Cervical biopsy
- HPV-positive patients - Echinacea (Active Comparator)
  Interventions: Diagnostic Test: Cervical biopsy
- HPV-positive patients - Standard (No Intervention)

INTERVENTIONS:
Diagnostic Test: Cervical biopsy — in office Cervical biopsy
  Arms: HPV-positive patients; HPV-positive patients - Echinacea

SUMMARY:
HPV is known to be the causal agent in the majority of cervical cancers. However, the role of the cervical bacterial microbiome in cervical cancer is not clear

ELIGIBILITY:
Inclusion Criteria:

* Women in fertile age

Exclusion Criteria:

* severe comorbidities

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Cervical microbiome | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Woman, Child and General and Specialized Surgery, University of Campania "Luigi Vanvitelli", Napoli, Italy

IPD SHARING:
Plan to Share IPD: No